CLINICAL TRIAL: NCT06239779
Title: Effects of Fibromyalgia Education on Smart Phone Addiction, Pain, and Quality of Life in Fibromyalgia Patients: A Randomized Controlled Study
Brief Title: Effects of Fibromyalgia Education on Smart Phone Addiction, Pain, and Quality of Life
Acronym: EFESAPQL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Selkin Yılmaz Muluk, MD, Physical Therapy and Rehabilitation specialist, Antalya Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Antalya AtatürkStateHospital
Record Dates: First submitted 2024-01-26; First posted 2024-02-02 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Fibromyalgia; Pain Syndrome; Addiction, Mobile Phone
Keywords: fibromyalgia; education; pain; phone addiction
MeSH Terms: conditions — Fibromyalgia; Somatoform Disorders; Technology Addiction; Pain | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled trial with a pre-post intervention (education) evaluation.
Who Masked: Participant, Investigator
Masking Description: In this study, both participant and investigator masking will be implemented to minimize potential bias and maintain objectivity. Participants in the education group will be unaware of the existence of the control group, and conversely, participants in the control group will be unaware of the education group. Additionally, to further ensure objectivity, after data collection, a secretary will anonymize patients into groups A and B using stickers. This comprehensive masking approach will prevent both participants and the investigator from being influenced by knowledge of group assignments during data analysis and interpretation, thereby enhancing research integrity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education Group (Experimental): The Education Group will be comprised of study participants who will receive an educational intervention aimed at enhancing their understanding and management of fibromyalgia. This group is designed to assess the impact of fibromyalgia education on various aspects of participants' well-being, including pain levels, smart phone addiction, and daily activities.
  Participants in the Education Group will attend an educational session. The educational content will cover the following key topics: an overview of fibromyalgia, coping strategies and potential harmful effects of smart phone addiction on fibromyalgia.
  The primary objective of the Education Group is to evaluate the influence of fibromyalgia education on pain levels, quality of life and physical function (measured using the FIQR) and smart phone addiction (measured using the SAS-SV), exercise frequency and daily screen time based on participant diaries.
  Interventions: Other: Education
- Control Group (No Intervention): The Control Group is a vital component of this study, serving as a reference group for evaluating the impact of the Education Group's intervention. Participants in this group will not receive the structured educational intervention. Instead they will follow their usual routines and receive standard care for fibromyalgia, which may include any recommendations typically offered by their healthcare providers but they are monitored similarly to the participants in the Education Group.
  The primary objective of the Control Group is to provide a baseline against which the effects of the educational intervention received by the Education Group can be compared. By not receiving the intervention, this group will help assess whether the educational program has a measurable impact on various aspects of participants' well-being when compared to standard care.

INTERVENTIONS:
Other: Education — The education intervention will involve a PowerPoint presentation delivered individually by a physician to each participant in intervention group, covering an overview of fibromyalgia, coping strategies, and the potential impact of smart phone addiction on fibromyalgia.
  Arms: Education Group

SUMMARY:
The study focuses on fibromyalgia, a condition characterized by chronic pain, fatigue, and associated issues like sleep disorders, depression, and anxiety. The investigators' goal is to detect smart phone addiction among fibromyalgia patients and assess potential decreases in pain and smart phone addiction after receiving fibromyalgia education.

Participants will report their recent exercise and screen time for the past week. They will also complete the Revised Fibromyalgia Impact Questionnaire (FIQR) to measure pain and physical function and the Smart Phone Addiction Scale-Short Version (SAS-SV) to assess smart phone use. Diaries will track daily exercise and screen time for 20 days.

The intervention group will receive fibromyalgia education, covering an overview of fibromyalgia, coping strategies, and discussions on the impact of digital addictions. This education, delivered via Microsoft PowerPoint program presentation by a physician, aims to help patients.

After 20 days, all participants will redo the FIQR and SAS-SV assessments, and diary data will be collected.

This study examines how physician-provided fibromyalgia education affects pain levels, smart phone addiction, exercise and screen times. The results will deepen our understanding of how education can enhance the lives of fibromyalgia patients and aid in developing more effective strategies to manage pain and improve their quality of life.

DETAILED DESCRIPTION:
Fibromyalgia is a musculoskeletal disease characterized by chronic pain, fatigue, and often accompanied by sleep disorders, depression, and anxiety. This study aims to identify smart phone addiction among fibromyalgia patients and explore potential improvements in their pain and smart phone addiction after receiving fibromyalgia education.

On the first day, all participants will be asked about their recent exercise duration and average screen time over the past week. They will then complete the FIQR to assess pain, quality of life and physical function in fibromyalgia, as well as the SAS-SV to measure smart phone use. Participants will receive their SAS-SV scores and be provided with diaries to record daily exercise and smart phone screen time for the next 20 days.

Patients in the intervention group will receive fibromyalgia education, which includes an overview of fibromyalgia, coping strategies (exercise, sleep management, stress reduction), and discussions on the impact of digital addictions like smart phone addiction on quality of life and stress levels. This education, presented as a face-to-face individual based Microsoft PowerPoint slide show, will be delivered by the researcher physician.

At the 20th-day follow-up, all participants will again complete the FIQR questionnaire and SAS-SV scale, and data from their diaries will be collected for further analysis.

This study aims to assess how fibromyalgia education provided by a physician affects pain levels, smart phone addiction (measured by FIQR and SAS-SV), exercise frequency, and daily screen time based on patient diaries. The findings will contribute to our understanding of how brief fibromyalgia education may impact the daily lives of patients and help develop more effective strategies to alleviate pain and enhance the quality of life for individuals with fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Fibromyalgia: Participants must have received a definitive diagnosis of fibromyalgia from a specialist. This diagnosis should have been made within the last 6 -months or they should be newly diagnosed with fibromyalgia.
* Ownership of a Smart Phone: Participants are required to own a smart phone as this is essential for aspects of the research related to smart phone addiction.
* Ability to Collaborate: Participants must be willing to actively participate in the research process, follow data collection procedures, and collaborate with the research team.

Exclusion Criteria:

* Cognitive Impairment or Severe Neurological/Psychiatric Illness: Individuals with significant cognitive impairment or severe neurological or psychiatric conditions that may affect their participation are excluded.
* Serious Health Conditions: Individuals with severe health conditions (e.g., cancer, chronic heart disease) that substantially affect their daily life and could confound the study outcomes are excluded.
* Other Addictions: Individuals with other types of addictions (e.g., alcohol, substance addiction) are not eligible for participation.
* Recent Serious Surgery or Trauma: Individuals who have undergone major surgery or experienced significant trauma recently are excluded.
* Unwillingness to Participate: Individuals who are unwilling to participate in the research process or who do not consent to be part of the study are excluded.
* Non-Compliance with Procedures: Individuals who are unable or unwilling to comply with data collection procedures as outlined by the research team are excluded.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2024-01-19 (Actual); Primary Completion 2024-06-19 (Actual); Study Completion 2024-06-24 (Actual)

PRIMARY OUTCOMES:
Pain Levels, Quality of Life, and Physical Function | This assessment is conducted at the beginning of the study (first day) and at the end of the study (20th day). Therefore, the time frame for this assessment spans from the first day to the 20th day of the study.
  These are measured using the Fibromyalgia Impact Questionnaire - Revised Form is a widely recognized instrument for assessing the impact of fibromyalgia on patients' lives. FIQR encompasses various dimensions, including pain levels, quality of life, and physical function. It employs a scale with a minimum value of 0, a maximum value of 100, and higher scores indicating worse outcome fibromyalgia impact. The study aims to assess the impact of fibromyalgia education on pain levels, quality of life, and physical function using this questionnaire.
Smart Phone Addiction | This assessment is conducted at the beginning of the study (first day) and at the end of the study (20th day). Therefore, the time frame for this assessment spans from the first day to the 20th day of the study
  This is measured using the Smartphone Addiction Scale-short version. The study aims to assess the impact of fibromyalgia education on smart phone addiction using this scale.

SECONDARY OUTCOMES:
Exercise Frequency | Participants start filling out the diary on the first day of the study and continue to do so every day for the entire 20-day duration of the study. The time frame for the diary entries covers the entire 20-day period.
  This outcome is evaluated based on participant diaries. The study intends to determine how fibromyalgia education may affect participants' exercise habits.
Daily Screen Time | Participants start filling out the diary on the first day of the study and continue to do so every day for the entire 20-day duration of the study. The time frame for the diary entries covers the entire 20-day period.
  This outcome is evaluated based on participants' self-reported daily screen time, retrieved from the settings of their smartphones and recorded in their diaries. The study intends to determine how fibromyalgia education may affect participants' daily screen time on smart phone.

CONTACTS AND LOCATIONS:
Overall Officials: Nazlı Ölçücü, MD, Study Director — Physical Medicine and Rehabilitation specialist; Selkin Yılmaz Muluk, MD, Principal Investigator — Antalya Ataturk State Hospital
Locations (1):
- Ataturk State Hospital, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The investigators do not plan to share questionnaires, scales, or patient diaries as they include personal data but are open to sharing the results of the data and the statistic analysis details upon reasonable request,
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Sharing will occur from the date of publication and continue for a period of three months thereafter.
Access Criteria: Access will be granted to researchers, institutions, or organizations with a legitimate research purpose directly related to the subject matter of the shared data. All parties seeking access must sign an agreement confirming their commitment to maintaining the confidentiality of the data and using it only for research purposes.

REFERENCES:
- [Background] Arnold LM, Bennett RM, Crofford LJ, Dean LE, Clauw DJ, Goldenberg DL, Fitzcharles MA, Paiva ES, Staud R, Sarzi-Puttini P, Buskila D, Macfarlane GJ. AAPT Diagnostic Criteria for Fibromyalgia. J Pain. 2019 Jun;20(6):611-628. doi: 10.1016/j.jpain.2018.10.008. Epub 2018 Nov 16. PMID 30453109
- [Background] Winslow BT, Vandal C, Dang L. Fibromyalgia: Diagnosis and Management. Am Fam Physician. 2023 Feb;107(2):137-144. PMID 36791450
- [Background] Nikolic A, Bukurov B, Kocic I, Vukovic M, Ladjevic N, Vrhovac M, Pavlovic Z, Grujicic J, Kisic D, Sipetic S. Smartphone addiction, sleep quality, depression, anxiety, and stress among medical students. Front Public Health. 2023 Sep 6;11:1252371. doi: 10.3389/fpubh.2023.1252371. eCollection 2023. PMID 37744504
- [Background] Kulekcioglu S, Cetin A. Social media use in patients with fibromyalgia and its effect on symptom severity and sleep quality. Adv Rheumatol. 2021 Aug 23;61(1):51. doi: 10.1186/s42358-021-00210-7. PMID 34425915